CLINICAL TRIAL: NCT01546818
Title: A Phase I, Randomized, Observer-blinded, Placebo-controlled Clinical Study to Assess the Safety, Tolerability, and Immune Response of Killed-Whole HIV-1 Vaccine (SAV001-H) Administered Intramuscularly to Chronic HIV-1 Infected Patients Currently Under Treatment With Highly Active Antiretroviral Therapy (HAART)
Brief Title: Safety and Immune Response Assessment Study of Killed-whole HIV-1 Vaccine (SAV001-H) in Chronic HIV-1 Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumagen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: SAV-CT01
Record Dates: First submitted 2009-06-09; First posted 2012-03-07 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-09

CONDITIONS: HIV Infections
Keywords: HIV; Vaccine; HIV-1 infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: SAV001-H — A whole-killed HIV

SUMMARY:
The purpose of this study is to examine the safety, tolerability, and immune response to killed-whole HIV-1 (SAV001-H) vaccine as a primary vaccination regimen in HIV infected individuals.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* Chronic HIV infection as defined by documentation of HIV infection for over ne year.
* Prior antiretroviral therapy defined as a minimum of 6 months of treatment with HAART. (HAART is defined as a combination of at least 2 antiretroviral agents.)
* CD4+ cell count more than 350 cells per mm3 for a period of 6 months prior to study entry at least at 3 different time points (one of which must be obtained at screening) obtained at any laboratory that possesses a CLIA certification or its equivalent.
* HIV-1 RNA levels less than 50 copies per mL for a period of 6 months prior to study entry at least at 3 different time points (one of which must be obtained at screening) by any laboratory that possesses a CLIA certification or its equivalent.
* Laboratory values obtained within 28 days prior to study entry
* Men and women between 18 and 50 years of age
* Female study volunteers of reproductive potential (defined as girls who have reached menarche or women who have not been post-menopausal for at least 24 consecutive months, i.e. who have had menses within the preceding 24 months, or have not undergone surgical sterilization (e.g. hysterectomy, bilateral oophorectomy, or salpingotomy) must have a negative serum or urine pregnancy test performed within 3 days before initiating study-specified medication.

If participating in sexual activity that could lead to pregnancy, the female study volunteer must use a form of contraception listed below while receiving protocol-specified medication and for 6 months after stopping the medication. At least one of the following methods MUST be used appropriately (with or without hormone-based method):

* Condoms (male or female) with or without a spermicidal agent
* Diaphragm or cervical cap with spermicide
* IUD

  * Informed of, and willing and able to comply with, the investigational nature of the study, and have signed an informed consent form in accordance with institutional and regulatory guidelines

Exclusion Criteria:

* History of serious adverse reactions to vaccines including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain, except for subjects who have a history of an adverse reaction to pertussis vaccine as a child may enroll.
* History of CD4+ counts less than 350 cells per mm3, opportunistic infections, or AIDS-defining illnesses.
* History of autoimmune disease, immunodeficiency (other than HIV infection), asthma, diabetes (including Type II diabetes or insulin resistance) requiring insulin or oral hypoglycemics, thyroid disease, bleeding disorder, active malignancy, viral hepatitis, or asplenia.
* HBVsAg, HCV Ab, or RPR positive.
* Suspected allergy or adverse reaction to any components of the study agent.
* Changes in antiretroviral regimen within 6 months prior to entry due to virologic failure (not including toxicities).
* Pregnancy or breast-feeding.
* Receipt of live attenuated vaccines or investigational research agents within 30 days prior to study entry.
* Receipt of blood products within 120 days prior to study entry.
* Receipt of immunoglobulin within 60 days prior to study entry.
* Receipt of medically indicated subunit or killed vaccines (e.g., influenza, pneumococcal, or allergy treatment with antigen injections) within 14 days prior to study entry.
* Receipt of prior experimental HIV vaccines.
* Any investigational antiretroviral agents that are not obtained through expanded access.
* Receipt of immunosuppressive medications within the past 6 months (e.g., oral/parenteral/inhaled corticosteroids, and/or cytotoxic medications). NOTE: The following will be allowed: corticosteroid nasal spray for allergic rhinitis; topical corticosteroids for acute, uncomplicated dermatitis; over the counter medications for acute, uncomplicated dermatitis for a period not longer than 14 days.
* Current anti-TB prophylaxis or therapy.
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.
* Serious illness (requiring systemic treatment and/or hospitalization) until subject either completes therapy or is clinically stable on therapy, in the opinion of the investigator, for at least 14 days prior to study entry.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2012-03; Primary Completion 2013-03 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Occurrence of at least one Grade 3 or higher adverse event, including signs/symptoms, lab toxicities, and/or clinical events possibly or definitely related to study treatment | 12 months

SECONDARY OUTCOMES:
To evaluate the immune response of killed-whole HIV-1 (SAV001-H) administered intramuscularly in individuals with chronic HIV-1 infection on HAART | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anthony M Mills, M.D., Principal Investigator — Anthony Mills MD Inc; Stefan Schneider, M.D., Principal Investigator — Living Hope Clinical Foundation
Locations (1):
- Anthony Mills, MD Internal Medicine, Los Angeles, California, United States